CLINICAL TRIAL: NCT06258226
Title: A Randomized Controlled Trial of Auricular Acupressure on Reduction of Estazolam in Patients With Insomnia
Brief Title: A Randomized Controlled Trial of Auricular Acupressure in Treating Estazolam-dependent Insomnia
Acronym: ESAAEDI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Qiqi Wu, Resident physician of TCM, Wenzhou Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y2023213
Record Dates: First submitted 2024-02-05; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Estazolam-dependent Insomnia
Keywords: auricular acupressure; estazolam; insomnia; drug-dependent; estazolam-dependent insomnia; randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional dosage reduction group (Active Comparator): The drug reduction method of estazolam tablets (Shanghai Xinyi Pharmaceutical Co., Ltd., Shanghai, China, State Drugs Administration License No.: H31020644, 1 mg) will be given, with a starting dose of 1 mg, that is, the dosage of estazolam will be reduced by 25% (0.25mg) every week until the dosage will be stopped completely on the premise of no aggravation of insomnia symptoms.
  Interventions: Drug: Conventional dosage reduction
- Auricular acupressure group (Experimental): Auricular acupressure therapy will be added based on the estazolam reduction method in the control group. The specific auricular points to be treated are Shenmen (TF4), Sympathetic (AH6), Endocrine (CO18), Heart (CO15), Liver (CO12) and Kidney (CO10). During the treatment, the acupuncturist will use a metal probe to identify the auricular points and ask the patients if they experience "deqi" sensations such as heat, numbness, distension, or pain. Once the auricular points have been confirmed, the ear will be disinfected using a 75% ethanol solution and dried using a sterile dry cotton ball. The acupuncturist will then hold the ear in place with their left hand while using their right hand to manipulate a tweezer and apply tape (0.5 x 0.5 cm) with vaccaria (Suzhou Konakang Medical Instrument Co., LTD., Suzhou, China) to the selected auricular point.
  Interventions: Procedure: Auricular acupressure
- Sham auricular acupressure group (Sham Comparator): Based on the estazolam reduction method in the control group, the acupuncturist will place the same skin-colored adhesive tapes without vaccaria on the auricular points, but these tapes will not be pressed during treatment.
  Interventions: Procedure: Sham auricular acupressure

INTERVENTIONS:
Drug: Conventional dosage reduction — The doctor will guide patients to adjust medication dosage once a week in the outpatient clinic. When patients experience withdrawal reactions such as worsening insomnia or anxiety symptoms due to drug reduction, they will be returned to the oral dose before the current reduction, and the dosage will be reduced again after evaluation in the next reduction cycle. The treatment for 4 weeks is one course and 1 course of treatment is required totally.
  Other Names: Estazolam reduction
  Arms: Conventional dosage reduction group
Procedure: Auricular acupressure — Auricular acupressure is a non-pharmacological therapy that involves applying acupressure on the surface of points in different parts of the ear. One side of the auricular acupoints will be treated first and the tapes will be kept in place for 3 days. On the fourth day, the tapes on the ear will be removed and new tapes will be applied to the opposite side of the ear. The purpose of replacing tapes is to reduce the adverse events (AEs) that may be caused by long-term stimulation unilaterally. In addition, the participants will be informed to press the tapes by themselves for 3 to 5 minutes vertically and appropriately to achieve the sensation, with a duration of 4 to 5 times a day. The treatment will last for 4 weeks, and the follow-up will be done after 1 month.
  Arms: Auricular acupressure group
Procedure: Sham auricular acupressure — Based on the estazolam reduction method in the control group, the acupuncturist will place the same skin-colored adhesive tapes without vaccaria on the auricular points, but these tapes will not be pressed during treatment.
  Arms: Sham auricular acupressure group

SUMMARY:
Insomnia is a disorder characterized by difficulties in falling asleep, maintaining sleep or waking up too early, and impairment of daytime functioning. Drug-dependent insomnia refers to insomnia patients taking sedatives and sleeping pills regularly for a long period of time, and becoming psychologically and physiologically dependent on them. In many countries, auricular acupressure (AA) has attracted growing attention as a complementary or alternative treatment for insomnia; however, there is a lack of rigorous randomized, controlled studies evaluating AA specifically for estazolam-dependent insomnia. Our proposed trial aims to assess the therapeutic effect of AA on estazolam-dependent insomnia.

DETAILED DESCRIPTION:
This study is a randomized, single-blinded, three-arm controlled trial. No less than 120 participants will be randomized into one of three groups: AA group, sham auricular acupressure (SAA) group, and conventional dosage reduction group. All treatments will be administered for 4 weeks, with a follow-up period of 1 month. The primary clinical outcomes will be estazolam dosing and reduction rates, serum gamma-aminobutyric acid (GABA) and cortisol (CORT) levels. Secondary outcomes will concern the Pittsburgh sleep quality index (PSQI) and Benzodiazepine Withdrawal Symptom Questionnaire (BWSQ). Both intention-to-treat and per-protocol analyses will be performed, with significance level determined as 5%.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for insomnia;
* Meet the diagnostic criteria for hypnotic drug-dependent insomnia;
* Regularly taking estazolam tablets for more than 2 months, and need to stop the medication;
* The dependent dosage of estazolam is 1mg, and withdrawal reaction occurs when the dosage is less than 1mg;
* PSQI score ≥ 7 (defined as "poor sleep quality", PSQI ≥ 7 is used as the reference threshold for judging sleep quality problems);
* Sign the informed consent.

Exclusion Criteria:

* Patients with cognitive disorders caused by cerebrovascular diseases, psychiatric disorders, and so on;
* Patients with serious heart, liver, kidney and blood system diseases;
* Patients with psychiatric illness/drug abuse (including alcohol);
* Patients who cannot cooperate with treatment, observation and evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Estazolam Dosing and Reduction Rates | Estazolam dosing will be assessed before treatment，1, 2, 3, and 4 weeks after treatment，1 month after follow-up visiting. The rate of dosage reduction will be observed 4weeks after treatment，1 month after follow-up visiting
  The amount of drug taken by patients will be assessed.The rate of dosage reduction will be observed. Estazolam reduction rate = (pre-treatment Estazolam dose - post-treatment Estazolam dose)/pre-treatment Estazolam dose x 100%.
Serum Gamma-aminobutyric acid and Cortisol Levels | Venous blood samples will be drawn twice from each patient at 8:00-9:00 in the morning 1 day before treatment and 1 day after the end of treatment.
  The method of enzyme-linked immunosorbent assay (ELISA) will be used. 4 ml of venous blood will be extracted from the subjects, and will be added anticoagulant. After that, the samples will be centrifuged at 3000 r/min to separate upper serum and preserved in a refrigerator at -80℃, according to the kit instructions.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline, 4 weeks after treatment commencement, and the 1-month follow-up
  The Pittsburgh Sleep Quality Index is a self-rated questionnaire used to assess sleep quality and disturbances over a 1-month period. It comprises 19 self-rated items and five other-rated items. The scores for the 19 self-rated items and five other-rated items are not included in the total score. Except for the first item, the remaining 18 items include the seven following subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficacy, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each subscale is rated from 0 to 3, and the accumulated scores of the seven subscales constitute the total score of the PSQI (0-21), where 7 is the threshold value of the sleep quality problem. A higher score indicates more severe sleep disorders.
Benzodiazepine Withdrawal Symptom Questionnaire | Baseline, 4 weeks after treatment commencement, and the 1-month follow-up
  A self-report questionnaire is described which records the main symptoms experienced during withdrawal from benzodiazepines in pharmacologically dependent patients. The questionnaire consists of 20 items

CONTACTS AND LOCATIONS:
Overall Officials: Qiqi Wu, Principal Investigator — Wenzhou Central Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu Q, Wang J, Fan L, Qian L, Han D, Hu H, Gao H. Efficacy and safety of auricular acupressure on reduction of estazolam in patients with insomnia: a study protocol for a three-arm, blinded randomized controlled trial. BMC Complement Med Ther. 2024 Oct 12;24(1):367. doi: 10.1186/s12906-024-04651-7. PMID 39395964